CLINICAL TRIAL: NCT04977349
Title: Manual Therapy Effectivity Combinated or Lonely With an Exercises Program for a Wind Musicians With Orofacial Pain
Brief Title: Manual Therapy Effectivity and Exercises in Musicians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Daniel Pecos Martín (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Daniel Pecos Martín, Vice-dean of Physiotherapy, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/40
Record Dates: First submitted 2020-12-01; First posted 2021-07-26 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Orofacial Pain
Keywords: Orofacial pain; Wind musicians; Manual Therapy; Exercise program
MeSH Terms: conditions — Facial Pain | interventions — Musculoskeletal Manipulations; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wind Musicians (Experimental): Isometric exercises for: cranial protrusion, mouth opening, laterality cervical movement and cervical coordination by laser assesment. And the manual therapy from the Active Comparator group.
  Interventions: Other: Manual Therapy; Other: Exercise program
- Wind musicians (Active Comparator): This group will be treated by manual therapy: suboccipital inhibition, myofascial extracavitary treatment in (superior trapezius fibers, Sternocleidomastoid (ECOM), masseter and temporalis) and intracavitary muscles (medialis and lateral pterygoid muscles).
  Interventions: Other: Manual Therapy; Other: Exercise program

INTERVENTIONS:
Other: Manual Therapy — This group will be treated by manual therapy: suboccipital inhibition, myofascial extracavitary treatment in (superior trapezius fibers, ECOM, masseter and temporalis) and intracavitary muscles (medialis and lateral pterygoid muscles).
Other: Exercise program — Isometric exercises for: cranial protrusion, mouth opening, laterality cervical movement and cervical coordination by laser assessment. And the manual therapy from the Active Comparator group.

SUMMARY:
Orofacial pain is one of the most common dysfunctions among wind musicians, a population with a high incidence of temporomandibular disorder (TMD). Regarding the treatment of TMD, the efficacy of manual therapy and therapeutic exercise has been studied, but there is a lack of high quality research supporting its implementation. There is, however, an agreement on the need of combining the treatment of the temporomandibular joint and the cervical spine, due to their close biomechanical relation.

Aims of the study: To analyse the efficacy of an evidence-based manual therapy protocol alone or in combination with an exercise program on the treatment of orofacial pain during musical practice on wind musicians. Furthermore, this study aims at observing whether if said treatment is more effective in the short, medium, or long term, and which variables are the most influenced.

DETAILED DESCRIPTION:
Methods: A sample of 40 wind musicians with orofacial pain during practice with the instrument will be recruited in the different conservatories of the Community of Madrid. The sample will be divided into two different groups: a control group who will receive the manual therapy protocol, and an experimental group who will, in addition, receive an exercise program. Treatment will consist of ten session distributed along 5 weeks, of an approximated duration of 30 minutes per session. Assessments will be carried out pre- and post-intervention, and for a two- and four-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Metal or wood wind musicians
* Orofacial pain during the practice in the last 30 days.
* More than 20 hours by week in the practice.
* Between 18-65 years old.

Exclusion Criteria:

* Neurological diseases.
* Analgesics previous treatments.
* Any trauma or bone fractures in skull or cervical spine.
* Any surgical intervention in cervical spine, orofacial region or temporo-mandibular joint.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Orofacial pain | Change from baseline at 2 months
  Visual Analogic Scale.The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured from 0 (no pain) to 10 (maximum pain). All the subjects will showed their pain level.
Pressure Pain Threshold | Change from baseline at 2 months
  An algometer Wagner FPI 10-WA will be used to determine the Pressure Pain Threshold in trigger points.
Range of Temporo mandibular Movement | Change from baseline at 2 months
  A vernier caliper will be used to measure mandibular movements. A vernier caliper is a validated tool to measure the opening, protusion, laterotrusion and overjet movements of the temporo mandibular joint
cervical range of movement (CROM) | Change from baseline at 2 months
  The instruments used to assess CROM will be a CROM goniometer. The CROM goniometer is a validated tool to measure the flexion, extension, rotation and tilt movements of the cervical spine.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Overall Study Officials, Alcalá de Henares, Madrid
  - Nursing and Physiotherapy Faculty, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No